CLINICAL TRIAL: NCT06729359
Title: Polycystic Ovary Syndrome and Urinary Tract Stones: a BMI-Adjusted Analysis in Iraqi Women
Status: Completed | Type: Observational
Sponsor: Al-Kindy College of Medicine (Other)
Responsible Party: Principal Investigator, Harth Mohamed Kamber, Assistant proffessor, Consultant utologist, Al-Kindy College of Medicine
Other Study IDs: 19 Al-KindyCM
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: PCOS (Polycystic Ovary Syndrome); Stone, Urinary; BMI; Obesity; Overweight; Underweight
Keywords: PCOS (Polycystic Ovary Syndrome); stone, urinary; BMI; Obesity; Overweight; Underweight
MeSH Terms: conditions — Polycystic Ovary Syndrome; Urinary Calculi; Obesity; Overweight; Thinness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PCOS (Polycystic Ovary Syndrome) group: includes patients diagnosed with PCOS (Polycystic Ovary Syndrome)
  Interventions: Diagnostic Test: Ultrasonography of the abdomen and pelvis
- Contorol group: include women of the same age group with no clinical or laboratory evidence of PCOS (Polycystic Ovary Syndrome)
  Interventions: Diagnostic Test: Ultrasonography of the abdomen and pelvis

INTERVENTIONS:
Diagnostic Test: Ultrasonography of the abdomen and pelvis — ultrasonography of the abdomen and pelvis using a 3.5mhz abdominal probe
  Other Names: tranveginal ultrasonography; serum testosterone; Serum dehydroepiandrosterone sulfate (DHEA-S); Serum androstenedione; Serum , luteinizing hormone (LH); Serum follicle-stimulating hormone (FSH); Serum sex hormone-binding globulin

SUMMARY:
The goal of this observational case-control study is to find out the impact of PCOS as a risk factor for the presence of urinary tract stones taking into account the BMI of women aged 18-40 years consulting the gynecology and obstetrics outpatient clinic at Al-Elwiya Maternity Teaching Hospital.

The study aims to collect information from approximately 200 women with polycystic ovary syndrome and 200 volunteers who do not have PCOS.

A written consent was obtained from all the participants. The information collected included age, weight, and height. In addition, focused history and clinical examination were conducted for all patients, and for some patients, one or more additional blood tests were obtained. The additional tests included but not limited to serum levels of testosterone, dehydroepiandrosterone sulfate (DHEA-S), androstenedione, luteinizing hormone (LH), follicle-stimulating hormone (FSH), and sex hormone-binding globulin. Moreover, ultrasonography of the abdomen and pelvis was obtained for all patients as part of the diagnosis of PCOS and as screening for urinary tract stones. Also, transvaginal ultrasonography was obtained for some patients according to the individual condition as requested by the treating gynecologist. The diagnosis ofc PCOS was based on the Rotterdam criteria. (1)

The main questions the study aims to answer are:

* Is PCOS a risk factor for urinary tract stones when taking BMI into account?
* Is PCOS a risk for urinary tract stones at all?
* Is there an association between PCOS and BMI?
* Does BMI affect the presence of urinary tract stones at all and the presence of urinary tract stones when taking PCOS into account?

ELIGIBILITY:
Inclusion Criteria:

* female
* age 18-40 years

Exclusion Criteria:

* A medical or surgical condition that affects urinary tract stone formation.
* A medical or surgical condition that affects body weight or height.
* A medical or surgical condition that affects hormonal balance.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: the study recruited two groups of females attending the gynecology and obstetrics outpatient clinic at Al-Elwiya Maternity Teaching Hospital. the first group contains women diagnosed with PCOS (Polycystic Ovary Syndrome) and the second group contains normal women attending the clinic for other causes that do not affect the body weight or the hormonal balance of the body
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
the association between PCOS (Polycystic Ovary Syndrome) and the presence of urinary tract stones controlled for BMI | at the time of enrollment

SECONDARY OUTCOMES:
the association between PCOS (Polycystic Ovary Syndrome) and BMI | at the time of enrollment
the association between BMI and the presence of urinary tract stones | at the time of enrollment
the association between BMI and the presence of urinary tract stones controlled for the presence of PCOS (Polycystic Ovary Syndrome) | at the time of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Harth Mohamed Kamber, FICMS (Uro.), Study Chair — University of Baghdad / Alkindy College of Medicine; Weqar Akram Hussein, FICMS (Gyn.), Principal Investigator — University of Baghdad / Alkindy College of Medicine; Zahraa Muhmmed Jameel Al-Sattam, FICMS (Gyn.), Principal Investigator — University of Baghdad / Alkindy College of Medicine; Kamal Al-Jawdah, MBChB, MRCS, FIBMS, Study Director — United Lincolnshire Teaching Hospitals NHS Trust
Locations (1):
- Al-Elwiya Maternity Teaching Hospital, Baghdad, Alrusafa, Iraq

IPD SHARING:
Plan to Share IPD: Undecided